CLINICAL TRIAL: NCT00459992
Title: Pilot Study of the Metabolic Effects of Betahistine Hydrochloride in Overweight Women
Brief Title: Effects of Betahistine Hydrochloride in Overweight Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 070126; 07-CH-0126
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2014-12-11

CONDITIONS: Obesity; Overweight; Overnutrition
Keywords: Obesity; Weight Gain; Adult; Histamine; Metabolism; Overweight
MeSH Terms: conditions — Obesity; Overweight; Overnutrition; Weight Gain | interventions — Betahistine

INTERVENTIONS:
Drug: Betahistine Hydrochloride

SUMMARY:
This study will evaluate the effects of a drug called betahistine on appetite and food intake in overweight women. Betahistine has been used for many years to treat vertigo (dizziness). It was taken off the market in the United States in 1970 because it was thought to be ineffective for vertigo, but is still used for this purpose in many other countries. Some research suggests that betahistine may reduce appetite and food intake.

Healthy overweight women between 18 and 50 years of age may be eligible for this study. Candidates must have a body mass index (BMI) between 30 and 40 and weigh less than 300 pounds. They are screened with a medical history and physical examination, blood and urine tests, electrocardiogram (EKG), breathing test and eating behavior questionnaires.

Participants are admitted to the NIH Clinical Center for a 3-day/2-night stay for the following procedures:

* Medication: Subjects take either betahistine (in one of three possible doses) or placebo capsules one time on the days of admission to the Clinical Center (day 1), three times on day 2 and two times on day 3.
* Blood tests and 24-hour urine collection.
* Resting metabolic rate: Subjects rest quietly for 1 hour after awakening and then rest again under a clear plastic hood or while wearing a face mask, breathing normally for about 25 minutes.
* DEXA scan to measure body fat, muscle, and bone mineral content: Subjects lie on a table above a source of X-rays while a very small dose of X-rays is passed through the body.
* Meal studies: Subjects food intake is measured on days 2 and 3.
* Questionnaires: Subjects complete questionnaires about how hungry or full they are feeling and rate how much they liked the foods they ate.

DETAILED DESCRIPTION:
Current medications for the long-term treatment of obesity are moderately effective at best. Therefore, research focusing on compounds that affect energy balance through novel mechanisms is warranted. Preliminary human and animal data suggest central nervous system histaminergic tone is important in the regulation of food intake. We therefore propose to study the effects of betahistine hydrochloride, a histamine analogue which has agonist activity at the histaminergic H1 receptor and antagonist/reverse agonist activity at the H3 receptor. Prior animal studies have suggested that betahistine suppresses food intake and reduces body weight, but there are sparse human data assessing the effects of betahistine on metabolism.

Betahistine s effects on women s food intake and metabolism will be evaluated through an inpatient randomized double-blind placebo controlled dose-ranging study. We will examine the acute effects of betahistine on food intake, hunger, and satiety, resting energy expenditure, and on hormones and substrates relevant for body weight regulation. If results suggest betahistine has salutary effects on food intake or metabolism in humans, these studies will lay the groundwork for additional investigations to assess the efficacy of betahistine in the treatment of obesity.

ELIGIBILITY:
* INCLUSION CRITERIA:

Volunteers will qualify if they meet the following criteria:

1. Good general health. In general, subjects will be required to take no medications. However, individuals taking medications for obesity-related co-morbid conditions, who have not had changes in dosage for more than 6 months, may be included, at the discretion of the principal investigator.
2. Age 18-50 years.
3. Female sex. In this pilot study, we seek to decrease the variability of subject response to the greatest extent possible. Since women have a higher prevalence of obesity than men, and tend to be the group that most uses weight loss pharmacotherapy, we will only study women in the pilot investigation. Subsequent studies with include both sexes.
4. Regular menses (either spontaneous or as a result of oral contraceptive pills) or post-menopausal status (no menses for at least 3 months).
5. Obesity, defined as body mass index (BMI) between 30 and 40 kg/m(2) but weight under 300 lbs, in order for subject to be able to undergo DEXA scanning with the Hologic instrument available in the Nuclear Medicine Department.
6. A negative pregnancy test at the initial evaluation. Sexually active women must be using an effective form of birth control. These methods include abstinence, oral contraceptives, an intrauterine device (IUD), levonogestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). (One of these methods must have been used by the subject for at least two months prior to the start of the study). If one of these cannot be used, contraceptive foam with a condom is recommended.
7. Willingness to participate in the research protocol.

   EXCLUSION CRITERIA:

   Volunteers will be excluded (and referred to non-experimental treatment programs as needed) for the following reasons:
   1. A presence of major illnesses: renal, hepatic (other than obesity-related steatosis), gastrointestinal, most endocrinologic (e.g., Cushing syndrome, hyper- or hypothyroidism, pheochromocytoma), hematological problems or pulmonary disorders; or porphyria;
   2. History of anaphylaxis, asthma, urticaria, rhinitis, allergic rash, or other allergic disease requiring antihistamine treatment; subjects with a history of antihistamine treatment for a self-limited allergic reaction such as to poison ivy or to a medication that they are no longer taking may be included at the discretion of the primary investigator.
   3. History of peptic ulcer disease;
   4. Baseline QT interval prolongation (greater than or equal to 480 msec QTc) because of reports of histaminergic compounds causing prolonged QT interval and cardiac arrhythmias in susceptible patients (i.e. those with prolonged QT interval at baseline);
   5. Current smokers of tobacco products;
   6. Self-reported lactose intolerance;
   7. Self-reported food allergy to foods used in standardized food array in this protocol or to betahistine itself;
   8. Subjects following a diet with specific food requirements such as vegetarian, vegan, or kosher because of the use of a standardized food array in this protocol;
   9. Subjects with a history of DSMIV classifiable eating disorders such as anorexia nervosa, bulimia nervosa, or binge-eating disorder will be excluded from the current proof-of-concept study;
   10. Women with reproductive potential who are pregnant or who are currently nursing an infant;
   11. Individuals who have current substance abuse or a psychiatric disorder or other condition that in the opinion of the investigators would impede competence or compliance or possibly hinder completion of the study;
   12. Subjects who regularly use prescription medications unrelated to the complications of obesity (especially vasoactive compounds such as calcium channel blockers, nitrates, beta-blockers, etc.), subjects using H2 blockers for dyspepsia, and subjects who require chronic use of antihistamines for allergic conditions; oral contraceptive use will be permitted, provided the contraceptive has been used for at least two months before starting study medication. The use of over-the-counter and prescription medications will be reviewed on a case-by-case basis; depending on the medication, subjects who have continued to take prescription medication for at least 3 months prior to study entry may be eligible. Allowable medications may include statins for the treatment of dyslipidemia and low-dose aspirin for primary prevention of acute coronary syndrome. Medications used for the treatment of hypertension will not be allowed because of the potential vasodilatory activity of betahistine.
   13. Recent (3 months) use of anorexiant medications;
   14. Weight change of more than 3% of body weight in the past two months;
   15. Subjects with a consistently (2 weeks apart) elevated systolic blood pressure of greater than 160 mm Hg and/or a diastolic blood pressure greater than 95 mm Hg.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-04-10; Primary Completion 2011-02-14 (Actual); Study Completion 2011-02-14 (Actual)

PRIMARY OUTCOMES:
Changes in food intake and appetite with betahistine treatment.

SECONDARY OUTCOMES:
Gut hormone assessment with betahistine treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Background] Vidal J. Updated review on the benefits of weight loss. Int J Obes Relat Metab Disord. 2002 Dec;26 Suppl 4:S25-8. doi: 10.1038/sj.ijo.0802215. PMID 12457296
- [Derived] Ballenger KL, Tugarinov N, Talvacchio SK, Knue MM, Dang Do AN, Ahlman MA, Reynolds JC, Yanovski JA, Marini JC. Osteogenesis Imperfecta: The Impact of Genotype and Clinical Phenotype on Adiposity and Resting Energy Expenditure. J Clin Endocrinol Metab. 2022 Jan 1;107(1):67-76. doi: 10.1210/clinem/dgab679. PMID 34519823
- [Derived] Ali AH, Yanoff LB, Stern EA, Akomeah A, Courville A, Kozlosky M, Brady SM, Calis KA, Reynolds JC, Crocker MK, Barak N, Yanovski JA. Acute effects of betahistine hydrochloride on food intake and appetite in obese women: a randomized, placebo-controlled trial. Am J Clin Nutr. 2010 Dec;92(6):1290-7. doi: 10.3945/ajcn.110.001586. Epub 2010 Sep 29. PMID 20881066